CLINICAL TRIAL: NCT00993876
Title: Cognitive Flexibility and Its Correlation to Sleep and Neuroplasticity In The Course Of Depression During Different Treatments
Brief Title: Cognitive Flexibility in Major Depression in the Course of Pharmacological and Psychotherapeutic Treatment
Acronym: Decoflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zentrum für Integrative Psychiatrie (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KO 2067
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Cognitive Performance in Major Depression
Keywords: Depression; CREB; cognitive performance; psychotherapy; SSRI; SNRI
MeSH Terms: conditions — Depression | interventions — Citalopram; Reboxetine; Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Selective serotonin reuptake inhibitor (SSRI) (Experimental): citalopram
  Interventions: Drug: citalopram
- Serotonin-norepinephrine reuptake inhibitor (SNRI) (Experimental): reboxetine
  Interventions: Drug: reboxetine
- IPT (Active Comparator): interpersonal psychotherapy
  Interventions: Behavioral: interpersonal psychotherapy

INTERVENTIONS:
Drug: citalopram — 20 to 30 mg per day for 4 weeks
  Arms: Selective serotonin reuptake inhibitor (SSRI)
Drug: reboxetine — 4 to 8 mg per day for 4 weeks
  Arms: Serotonin-norepinephrine reuptake inhibitor (SNRI)
Behavioral: interpersonal psychotherapy
  Arms: IPT

SUMMARY:
Cognitive deficits in major depression seem explicable by the well-recognized concept of impaired neuroplasticity in mood disorders. This concept initially emerged from preclinical evidence that antidepressants phosphorylate and therefore activate the cyclic AMP response element binding protein (CREB) that is essential for synaptic plasticity. Nevertheless, the question remains whether the activation of CREB by antidepressants is relevant for the remission of cognitive deficits in patients. We addressed this issue by investigating the cognitive improvement during treatment with either citalopram or reboxetine because these antidepressants are different in their capacity to increase phosphorylated CREB (pCREB). Besides the pharmacological treatment groups, another group of patients was treated exclusively with psychotherapy.

DETAILED DESCRIPTION:
We randomly assigned forty-five depressive patients to one of three treatment groups (Citalopram, Reboxetin or interpersonal psychotherapy (IPT)). At baseline, day 7 and day 28 we assessed the severity of depression and the cognitive performance with respect to cognitive flexibility, memory and attention. We measured pCREB with an enzyme linked immuno sorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed according DSM-IV criteria as suffering from major depressive disorder
* A baseline score of at least 18 in the Hamilton Depression Scale (HAMD)
* No psychopharmacological treatment at least one week prior inclusion or 3 days wash-out

Exclusion Criteria:

* Severe depressive episode and/or psychotic depressive episode

Axis I disorder:

* Substance-related Disorders
* Psychotic Disorders
* Dementia or other cognitive Disorders
* Obsessive-Compulsive Disorders

Axis II disorder:

• Borderline Personality Disorder

Axis III disorder:

* Infectious Diseases
* Cancer
* Endocrinological Diseases
* Hematological Diseases
* Autoimmune Diseases

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
cognitive performance with respect to cognitive flexibility, memory and attention | 4 weeks

SECONDARY OUTCOMES:
CREB-phosphorylation in T-Lymphocytes | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jakob M. Koch, M.D., Principal Investigator — Zentrum für Integrative Psychiatrie, Kiel, Germany
Locations (1):
- Zentrum für Integrative Psychiatrie, Kiel, Germany